CLINICAL TRIAL: NCT02954562
Title: Physiological Correlates of Anxiety Associated With a Life-threatening Illness.
Brief Title: Correlates of Anxiety Associated With a Life-threatening Illness
Status: Completed | Type: Observational
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: MDA1-S1
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Anxiety
Keywords: anxiety; fMRI; emotion regulation
MeSH Terms: conditions — Anxiety Disorders; Emotional Regulation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anxiety: Participants enrolled in study ""A randomized, Double-Blind, Placebo-Controlled Phase 2 Pilot Study of MDMA-Assisted Psychotherapy for Anxiety Associated with a Life-Threatening Illness" (NCT02427568)" who meet further inclusion criteria for fMRI scan
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — Participants will undergo two to three fMRI scans
  Other Names: Functional magnetic resonance imaging

SUMMARY:
The goal of this observational trial is to gather brain scan data on people undergoing MDMA-assisted therapy. The main question it aims to answer is:

-How does brain activity change while completing an emotional regulation task in participants receiving MDMA-assisted therapy?

Researchers will compare participants receiving MDMA-assisted therapy to participants receiving placebo plus therapy.

Participants will undergo baseline brain scans with functional magnetic imaging (fMRI) while they perform an emotional regulation task and other attentional tasks.

Participants will then undergo two medication sessions of MDMA or placebo-assisted therapy. Then, undergo another brain scan. Participants will then undergo a third medication session and repeat the brain scans.

DETAILED DESCRIPTION:
A subset of participants in the study "Randomized, Double-Blind, Placebo-Controlled Phase 2 Pilot Study of MDMA-Assisted Psychotherapy for Anxiety Associated with a Life-Threatening Illness" (NCT02427568) without any contraindicating factors for brain imaging will undergo three fMRI scans as part of this observational study. The first scan will occur prior to experimental sessions and a second scan will occur after two experimental sessions of MDMA or placebo-assisted psychotherapy. Participants will then be scanned a third time after they have completed a total of three sessions of MDMA-assisted psychotherapy (this includes both participants that are originally in the MDMA-assisted psychotherapy group, as well as the participants in the placebo group who will cross over and complete three active MDMA-assisted psychotherapy sessions subsequent to their placebo-assisted psychotherapy). The primary endpoint will be the scan after the second experimental session.

During each scanning session, participants will be undergoing brain scans with functional magnetic imaging (fMRI) while they perform an emotional regulation task that involves observing images with negative emotional valence. These images are drawn from, and have their emotional valence validated by, the International Affective Picture System (IAPS). Participants are instructed either to view passively or attempt to reduce the negative affect associated with the images. In addition, resting state brain scans will be acquired while participants fixate on a central cross with no explicit task. Heart rate variability will be measured during these resting state scans. The comparison of changes in brain activity during execution of the emotional regulation task (as compared to baseline scans) after receiving psychotherapy with MDMA or placebo, as well as comparison of changes in resting state functional connectivity, are the primary outcome measures. Study observations are intended to assess changes in response to emotion-provoking material at several levels, most notably brain activity in response to anxiety producing images.

While in the scanner, participants will also listen to prerecorded audio scripts about life stresses for themselves and for another person with instructions to practice compassion for themselves or for others. Participants will additionally perform an attentional bias task where they respond to a dot-probe that appears following a brief presentation of paired images known to produce positive and negative emotions as their brain activity is measured and their reaction times are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the parent study, "A randomized, Double-Blind, Placebo-Controlled Phase 2 Pilot Study of MDMA-Assisted Psychotherapy for Anxiety Associated with a Life-Threatening Illness" (NCT02427568)"

Exclusion Criteria:

* Have a brain mass or lesion
* Have metal in their skulls,
* Having brain or heart pacemakers
* History of major head trauma
* Have past or present panic or extreme discomfort with being in small enclosed spaces (claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who can safely undergo and are willing to have fMRI scans and who are enrolled in the study ""A randomized, Double-Blind, Placebo-Controlled Phase 2 Pilot Study of MDMA-Assisted Psychotherapy for Anxiety Associated with a Life-Threatening Illness" (NCT02427568)"
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2015-11-07 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in fMRI Blood Oxygen Level Dependent (BOLD) responses to emotional regulation task | Two months after enrollment in study NCT02427568)
  Changes in brain activity during passive observation versus attempts to reduce negative response to images
Changes in fMRI Blood Oxygen Level Dependent (BOLD) resting state functional connectivity | Two months after enrollment in study NCT02427568)
  Changes in brain activity during resting state fMRI

SECONDARY OUTCOMES:
Heart rate variability (HRV) during own versus other's anxiety script | Two months after enrollment in study NCT02427568)
  Measuring changes in speed of heart rate while listening to a personalized versus a non-personalized anxiety script.
Changes in fMRI BOLD response during dot probe task | Two months after enrollment in study NCT02427568)
  Assess response to images evoking positive or negative emotion
Response time to dot probe task | Two months after enrollment in study MDA-1
  Response time (RT) to viewing positive or negative valence images
Measure of compassion for self versus other | Two months after enrollment in study NCT02427568)
  Compassion response listening to self-generated versus other-generated scripts

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silver, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California - Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No